CLINICAL TRIAL: NCT01204437
Title: An Investigational Randomized Study on Epirubicin Plus Cyclophospamide (EC) or Cyclophosphamide Plus Methotrexat Plus 5-fluorouracil (CMF) Versus Nab-paclitaxel Plus Capecitabine as Adjuvant Chemotherapy for Elderly Non Frail Patients With an Increased Risk for Relapse of a Primary Carcinoma of the Breast
Brief Title: Adjuvant Chemotherapy for Elderly Non Frail Patients With an Increased Risk for Relapse of a Primary Carcinoma of the Breast
Acronym: ICE-II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 52; 2008-003995-23 (EudraCT Number)
Record Dates: First submitted 2010-09-10; First posted 2010-09-17 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: adjuvant chemotherapy; primary carcinoma; elderly non frail patients; EC; CMF; Capecitabine; Nab-Paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — EC regimen; Cyclophosphamide; Methotrexate; Fluorouracil; Capecitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EC standard chemotherapy 4 cycles (Active Comparator)
  Interventions: Drug: Epirubicin, Cyclophosphamide
- CMF standard chemotherapy 6 cycles (Active Comparator)
  Interventions: Drug: Cyclophosphamide, Methotrexate, 5 FU
- Nab-Paclitaxel + Capecitabine 6 cycles (Experimental): 6 cycles of weekly nab-Paclitaxel 100 mg/m2 on days 1, 8, 15 q22 with a week of rest every 6 weeks in combination with capecitabine 2000 mg/m2, days 1 - 14 orally, divided into 2 daily doses every 3 weeks for 6 cycles
  Interventions: Drug: Capecitabine, Nab-Paclitaxel

INTERVENTIONS:
Drug: Epirubicin, Cyclophosphamide — 4 cycles of chemotherapy with epirubicin plus cyclophosphamide (EC) on day 1 q22
  Arms: EC standard chemotherapy 4 cycles
Drug: Cyclophosphamide, Methotrexate, 5 FU — 6 cycles CMF on days 1 and 8 q29 Cyclophosphamide (500mg/qm), Methotrexate (40 mg/qm), 5 FU (600mg/qm)
  Arms: CMF standard chemotherapy 6 cycles
Drug: Capecitabine, Nab-Paclitaxel — 6 cycles of weekly nab-paclitaxel 100 mg/m2 on days 1, 8, 15 q22 with a week of rest every 6 weeks in combination with capecitabine 2000 mg/m2, days 1 - 14 orally, divided into 2 daily doses every 3 weeks for 6 cycles
  Arms: Nab-Paclitaxel + Capecitabine 6 cycles

SUMMARY:
Although approximately 50% of new diagnosis breast cancers are in patients above the age of 65, elderly people remain substantially under-represented in clinical trials, and therefore are under-treated. A recent trial of the CALBG in patient's ≥ 65 years with medium risk of breast cancer demonstrated an improved disease-free and overall survival for those treated with AC or CMF compared to those treated with capecitabine alone.

The primary aim of the ICE II trial is to determine the compliance and toxicity of epirubicin plus cyclophosphamide (EC) or CMF versus nab-paclitaxel plus capecitabine as adjuvant therapy in non frail elderly patients.

DETAILED DESCRIPTION:
Primary Objective:

Phase II:

To determine the compliance and safety of epirubicin plus cyclophosphamide or CMF (EC/CMF) and nab-paclitaxel in combination with capecitabine (PX).

Secondary Objective(s):

1. To compare the disease-free survival (DFS) and distant disease free survival (DDFS) with epirubicin plus cyclophosphamide or CMF (EC/CMF) vs. nab-paclitaxel in combination with capecitabine (PX).
2. To compare the overall survival (OS) with epirubicin plus cyclophosphamide or CMF (EC/CMF) vs nab-paclitaxel in combination with capecitabine (PX).
3. To analyze the efficacy of treatments in subgroups according to clinical stratification factors.
4. To determine prognostic factors on tumor tissue collected from primary surgery and to correlate them with study treatment effect.
5. To compare the geriatric assessments scores (Charlson, VES-13, IADL, G8) at baseline and end of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for all study procedures must be obtained and documented according to local regulatory requirements prior to beginning specific protocol procedures.
2. Complete baseline documentation must be sent to GBG Forschungs GmbH.
3. Histological confirmed unilateral or bilateral primary carcinoma of the breast.
4. Female and male breast cancer patients with age at first histologically diagnosis and axilla dissection ≥ 65 years.
5. Adequate surgical treatment with complete resection (R0) of the tumor and ≥ 10 axillary nodes. Sole sentinel node biopsy is allowed if the sentinel node shows no tumor involvement.
6. No evidence for distant metastasis at bone scan, liver ultrasound and chest x-ray.
7. Patients with stage pT3/4 or pN2/3 (≥ 4 involved lymph nodes) irrespective of additional risk factors.
8. Patients with stage pT1/2 and pN0/1 (0-3 involved lymph nodes) with an increased risk according to the clinico-pathological or uPA/PAI-1 criteria.
9. ECOG Performance Status <= 2.
10. Charlson Scale <= 2.
11. Estimated life expectancy of at least 5 years (irrespective of breast cancer diagnosis).
12. The patient must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre which could be the Principal or a Co- investigator's site.

Exclusion Criteria:

1. Known hypersensitivity reaction to the compounds or incorporated substances or known dihydropyrimidine dehydrogenase deficiency.
2. Low risk patient according to risk assessment.
3. Inadequate organ function including:

   Leucocytes < 3,5 G/l, Platelets < 100 G/l , Creatinine or Bilirubin above normal limits (1,25 above upper normal limit), Creatinine-Clearance below 50 ml/min, uncompensated cardiac function, severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study.
4. Previously or currently one of the following medical conditions:

   * pre-existing motor or sensory neuropathy of a severity >= grade 2 by NCI-CTC criteria;
   * history of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent;
   * known or suspected congestive heart failure (> NYHA I) and/or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, un- or poorly controlled arterial hypertension (i.e. BP >150/100 mmHg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease;
   * Creatinine Clearance less than 50 ml/min;
   * another primary malignancy with an event-free survival of < 5 years, except curatively treated basalioma of the skin and carcinoma in situ of the cervix.
5. Time since axillary dissection > 3 months.
6. Locally advanced, non-operable breast cancer.
7. Previous invasive breast carcinoma.
8. Prior chemotherapy for any malignancy.
9. Concurrent specific systemic anti-tumor treatment or treatment with experimental compounds within the last 6 months.
10. Concurrent treatment with other tumor specific experimental drugs. Participation in another clinical trial with any investigational not marketed drug.
11. Concurrent treatment with virostatic agents like sorivudine or analogues like brivudine, concurrent treatment with aminoglycosides, anticoagulants: heparin, warfarin as well as acetylic acid (e.g. Aspirin®) at a dose of > 325mg/day or clopidogrel at a dose of > 75 mg/day).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To determine the compliance and safety of epirubicin plus cyclophosphamide or CMF (EC/CMF) and nab-paclitaxel in combination with capecitabine (PX). | 4 months after Last Patient Out

SECONDARY OUTCOMES:
To compare the disease-free survival (DFS) and distant disease free survival (DDFS) with epirubicin plus cyclophosphamide or CMF (EC/CMF) vs. nab-paclitaxel in combination with capecitabine (PX). | After 4.5 years of Follow Up
To compare the overall survival (OS) with epirubicin plus cyclophosphamide or CMF (EC/CMF) vs nab-paclitaxel in combination with capecitabine (PX). | After 4.5 years of Follow Up
To analyze the efficacy of treatments in subgroups according to clinical stratification factors. | After 4.5 years of Follow Up
To determine prognostic factors on tumor tissue collected from primary surgery and to correlate them with study treatment effect. | After 4.5 years of Follow Up
To compare the geriatric assessment scores (Charlson, VES-13, IADL, G8) at baseline and end of therapy | 4 months after Last Patient Out

CONTACTS AND LOCATIONS:
Overall Officials: Gunter von Minckwitz, Prof., Principal Investigator — GBG Forschungs GmbH
Locations (1):
- German Breast Group, GBG Forschungs GmbH, Neu-Isenburg, Germany

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241